CLINICAL TRIAL: NCT03520413
Title: Practical Telemedicine to Improve Control and Engagement for Veterans With Clinic-Refractory Diabetes Mellitus (PRACTICE-DM)
Brief Title: Practical Telemedicine to Improve Control and Engagement for Veterans With Clinic-Refractory Diabetes Mellitus
Acronym: PRACTICE-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 16-213
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Telemedicine
Keywords: Complex Care; Outcomes; Telemedicine; Rural Health; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: VA Home Telehealth (HT) nurses will deliver the 5 intervention components during telephone encounters. The standard encounter frequency will be every two weeks, but may be extended to every 4 weeks for participants achieving their HbA1c goal. Should Veterans relapse while receiving the lower encounter frequency, HT will return to every-two-week encounters until the next HbA1c assessment. The 5 intervention components are: Telemonitoring, Self-management support, Diet/activity support, Medication management, & Depression support
Who Masked: Outcomes Assessor
Masking Description: Because participants will receive information on both study arms during the consent process, we will not attempt to blind participants to randomization assignment. However, in order to assure blinding of the staff that manage outcome data collection, randomization (including participant notification of group assignment by phone) will be managed by the project coordinator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRACTICE-DM (Experimental): PRACTICE-DM is a comprehensive telemedicine intervention that bundles telemonitoring, self-management support, diet/activity support, medication management, and depression support - each of which targets a critical factor underlying PPDM - into a single, comprehensive program specifically developed for practical delivery using existing VHA Home Telehealth (HT) workforce, infrastructure, and technical resources.
  Interventions: Other: PRACTICE-DM
- Standard VA Home Telehealth (Active Comparator): Standard VA HT care coordination and telemonitoring.
  Interventions: Other: Standard VA Home Telehealth

INTERVENTIONS:
Other: PRACTICE-DM — Five-component diabetes intervention: 1) telemonitoring; 2) self-management support; 3) diet/activity support; 4) medication management; and 5) depression support.
  Arms: PRACTICE-DM
Other: Standard VA Home Telehealth — Standard VA HT care coordination and telemonitoring.
  Arms: Standard VA Home Telehealth

SUMMARY:
Diabetes generates significant morbidity, mortality, and costs within the Veterans Health Administration (VHA). Veterans with persistently poor diabetes control despite clinic-based care are among the highest-risk diabetes patients in VHA, and contribute disproportionately to VHA's massive burden of diabetes complications and costs. VHA critically needs effective, practical management alternatives for Veterans whose diabetes does not respond to clinic-based management. The proposed study will address this need by leveraging VHA's unique Home Telehealth capacity to deliver comprehensive telemedicine-based management for Veterans with persistently poor diabetes control despite clinic-based care. Because this intensive intervention is delivered using only existing Home Telehealth workforce, infrastructure, and technical resources - which are ubiquitous at VHA centers nationwide - it could represent an effective, practical approach to improving outcomes in Veterans with PPDM, potentially translating to a substantial reduction in VHA's diabetes burden.

DETAILED DESCRIPTION:
This study will evaluate a comprehensive telemedicine intervention for Veterans with persistently poor diabetes control despite clinic-based Veterans Health Administration (VHA) care. Because this approach is designed for delivery via existing Home Telehealth (HT) services, which are ubiquitous throughout VHA, it may represent an effective, practical alternative for Veterans whose diabetes is refractory to clinic-based care.

Although efforts by clinicians and researchers have improved diabetes control across VHA, Veterans with persistent poorly-controlled diabetes mellitus (PPDM) have not benefitted from these advances. The investigators define PPDM as maintenance of a hemoglobin A1c (HbA1c) 8.5% for >1 year, despite receiving clinic-based diabetes care during this period. Veterans meeting this definition - approximately 12% of all Veterans with type 2 diabetes - contribute disproportionately to VHA's burden of diabetes complications and costs.

While clinic-based care is insufficiently effective in PPDM, telemedicine-based management that comprehensively addresses factors underlying poor diabetes control could improve outcomes for these high-risk Veterans. Unfortunately, healthcare systems have rarely integrated comprehensive telemedicine-based care into real-world practice, even for clinic-refractory conditions like PPDM. This gap stems from the fact that comprehensive telemedicine-based diabetes care has not previously been designed for practical delivery under real-world conditions. In order for telemedicine to fulfill its potential as a means to reduce the burden of PPDM, interventions must be developed with an emphasis on feasible delivery through existing workforce, infrastructure, and technical resources, such that effective implementation is eventually achievable. Until then, Veterans with PPDM will be left without alternatives when clinic-based care proves inadequate.

The proposed trial will evaluate Practical Telemedicine to Improve Control and Engagement for Veterans with Clinic-Refractory Diabetes Mellitus (PRACTICE-DM), a novel, comprehensive telemedicine intervention for PPDM that is designed for practical delivery within VHA. The Specific Aims of this study are to: 1) determine PRACTICE-DM's effectiveness; 2) evaluate PRACTICE-DM's acceptability and mechanisms of effect using a mixed method process evaluation; and 3) understand costs associated with PRACTICE-DM.

Two hundred Veterans with PPDM from two sites (Durham, North Carolina (NC) and Richmond, Virginia (VA)) will be randomized to receive one of two HT-delivered interventions: 1) PRACTICE-DM, a comprehensive intervention combining telemonitoring, self-management support, diet/activity support, medication management, and depression support; or 2) an active control, standard HT care coordination and telemonitoring. Both interventions will be delivered over a 12-month period and all participants will continue to receive usual VHA care.

The primary study outcome will be change in HbA1c from study baseline to 12 months. The secondary outcomes are guided by a theoretical framework, and will include diabetes self-care, diabetes burden, self-efficacy, and depressive symptoms. Qualitative interviews will be conducted with 20 intervention-group Veterans, the HT nurses delivering the intervention, and administrators at each site. Intervention costs will be comprehensively assessed and compared to standard HT care coordination and telemonitoring.

Although VHA is a leader in telemedicine, its telemedicine capabilities are currently underutilized for Veterans with PPDM. These Veterans are refractory to clinic-based care, so contribute disproportionately to diabetes complications and costs. This study will leverage VHA's unique telemedicine infrastructure to deliver comprehensive management designed for PPDM, with the goal of improving outcomes in this high-risk, high cost population. Because the proposed intervention is designed for delivery using existing HT services, it may represent an effective, practical approach to reducing the burden of poor diabetes control across VHA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with persistently poorly-controlled type 2 diabetes mellitus defined as the presence of 2 HbA1c values 8.5% during the prior year (none <8.5%) despite 1 or more appointments with a VHA Primary Care Provider (PCP) or Endocrinology during this period.

Exclusion Criteria:

* age >70
* life expectancy <5 years, or other comorbidities that would offset the benefits of HbA1c <8.5%
* inability to communicate by telephone
* dementia or psychosis
* active alcohol/substance disorder
* pregnancy
* prior hypoglycemic seizure/coma
* refusal to perform self-monitored blood glucose (SMBG)
* use of insulin infusion pumps
* hospitalized for stroke, heart attack or had surgery for blocked arteries in the past 12m
* receiving kidney dialysis
* metastatic cancer diagnosis
* use of a continuous blood glucose monitor (due to HT equipment constraints)
* primary provider requests patient not participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Crowley, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kobe EA, Edelman D, Tarkington PE, Bosworth HB, Maciejewski ML, Steinhauser K, Jeffreys AS, Coffman CJ, Smith VA, Strawbridge EM, Szabo ST, Desai S, Garrett MP, Wilmot TC, Marcano TJ, Overby DL, Tisdale GA, Durkee M, Bullard S, Dar MS, Mundy AC, Hiner J, Fredrickson SK, Majette Elliott NT, Howard T, Jeter DH, Danus S, Crowley MJ. Practical telehealth to improve control and engagement for patients with clinic-refractory diabetes mellitus (PRACTICE-DM): Protocol and baseline data for a randomized trial. Contemp Clin Trials. 2020 Nov;98:106157. doi: 10.1016/j.cct.2020.106157. Epub 2020 Sep 21. PMID 32971277
- [Result] Lewinski AA, Crowley MJ, Miller C, Bosworth HB, Jackson GL, Steinhauser K, White-Clark C, McCant F, Zullig LL. Applied Rapid Qualitative Analysis to Develop a Contextually Appropriate Intervention and Increase the Likelihood of Uptake. Med Care. 2021 Jun 1;59(Suppl 3):S242-S251. doi: 10.1097/MLR.0000000000001553. PMID 33976073
- [Result] Crowley MJ, Tarkington PE, Bosworth HB, Jeffreys AS, Coffman CJ, Maciejewski ML, Steinhauser K, Smith VA, Dar MS, Fredrickson SK, Mundy AC, Strawbridge EM, Marcano TJ, Overby DL, Majette Elliott NT, Danus S, Edelman D. Effect of a Comprehensive Telehealth Intervention vs Telemonitoring and Care Coordination in Patients With Persistently Poor Type 2 Diabetes Control: A Randomized Clinical Trial. JAMA Intern Med. 2022 Sep 1;182(9):943-952. doi: 10.1001/jamainternmed.2022.2947. PMID 35877092
- [Derived] Duffy RA, Jeffreys AS, Coffman CJ, Alexopoulos AS, Tarkington PE, Bosworth H, Edelman D, Crowley MJ. Evaluating Therapeutic Inertia in Two Telehealth Interventions for Type 2 Diabetes: Secondary Analyses of a Randomized Trial. Telemed J E Health. 2024 Jun;30(6):e1790-e1797. doi: 10.1089/tmj.2023.0453. Epub 2024 Feb 19. PMID 38377570

RESULTS

PARTICIPANT FLOW:
Groups:
- PRACTICE-DM: PRACTICE-DM is a comprehensive telemedicine intervention that bundles telemonitoring, self-management support, diet/activity support, medication management, and depression support - each of which targets a critical factor underlying Persistently Poorly controlled Diabetes Mellitus (PPDM) - into a single, comprehensive program specifically developed for practical delivery using existing Veterans Health Administration (VHA) Home Telehealth (HT) workforce, infrastructure, and technical resources.
  PRACTICE-DM: Five-component diabetes intervention: 1) telemonitoring; 2) self-management support; 3) diet/activity support; 4) medication management; and 5) depression support.
Period: Overall Study
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
Started | 101 | 99
Completed | 77 (Completed defined as Hemoglobin A1c collected at 12months) | 73 (Completed defined as Hemoglobin A1c collected at 12months)
Not Completed | 24 | 26
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 0 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Completed a study interview but did not obtain HbA1c data | 19 | 19

BASELINE CHARACTERISTICS:
Population: Randomized patients with persistently poorly controlled diabetes mellitus
Groups:
- Total: Total of all reporting groups
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 75 | 151
  >=65 years | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.3) | 57.8 (8.0) | 57.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 77 | 78 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 95 | 93 | 188
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 68 | 76 | 144
  White | 25 | 17 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Richmond, VA | 44 | 41 | 85
  United States: Durham, NC | 57 | 58 | 115
Baseline Hemoglobin A1c [Mean (Standard Deviation); unit: % HbA1c] | 10.1 (1.2) | 10.2 (1.4) | 10.2 (1.3)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (6.4) | 35.2 (7.0) | 34.8 (6.7)
Diabetes Distress Scale (DDS) [Mean (Standard Deviation); unit: units on a scale] — Scale 1-6. Higher score indicates higher distress level.
  units on a scale | 1.9 (0.7) | 1.9 (0.9) | 1.9 (0.8)
Diabetes Self-Management Questionnaire (DSMQ) [Mean (Standard Deviation); unit: units on a scale] — Scale 0-3. Scoring: Sum and transform to fall between 0-10. Higher score indicates more effective self-care.
  units on a scale | 6.9 (1.5) | 6.5 (1.7) | 6.7 (1.6)
Self-Efficacy (PCS) [Mean (Standard Deviation); unit: units on a scale] — Scale 1-7. Higher score indicates greater confidence.
  units on a scale | 5.2 (1.5) | 5.2 (1.4) | 5.2 (1.5)
Depression (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — Scale 0-3, Scoring average of responses 0-24. Higher score indicates greater depressive symptoms.
  units on a scale | 7.0 (5.2) | 7.6 (6.1) | 7.3 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Laboratory blood test to measure diabetes control
Time Frame: 12 months
Population: Mixed models were used to analyze outcomes. This methodology uses all observations from baseline and the follow-up timepoints. Therefore 200 observations were included at baseline and 150 observations at 12 months.
Measure: Mean (95% Confidence Interval); unit: % HbA1c
Groups:
- PRACTICE-DM: PRACTICE-DM is a comprehensive telemedicine intervention that bundles telemonitoring, self-management support, diet/activity support, medication management, and depression support - each of which targets a critical factor underlying Persistently Poorly controlled Diabetes Mellitus (PPDM) - into a single, comprehensive program specifically developed for practical delivery using existing VHA Home Telehealth (HT) workforce, infrastructure, and technical resources.
  PRACTICE-DM: Five-component diabetes intervention: 1) telemonitoring; 2) self-management support; 3) diet/activity support; 4) medication management; and 5) depression support.
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
Number analyzed (Participants) | 101 | 99
% HbA1c | 8.58 [8.22 to 8.94] | 9.19 [8.83 to 9.55]
Statistical Analysis 1: Comparison: PRACTICE-DM vs Standard VA Home Telehealth; Test type: Equivalence — Difference between groups at 12months; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.12 to -0.11]

2. Secondary Outcome: Diabetes Distress Scale
Description: Measure of diabetes distress and burden using the Diabetes Distress Scale (DDS). 17 items, Scale 1-6. Scoring: Average. Higher score indicates higher distress level.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
Number analyzed (Participants) | 101 | 99
score on a scale | 1.43 [1.30 to 1.56] | 1.67 [1.54 to 1.81]
Statistical Analysis 1: Comparison: PRACTICE-DM vs Standard VA Home Telehealth; Test type: Equivalence — Difference between groups at 12months; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.42 to -0.07]

3. Secondary Outcome: Diabetes Self-Management Questionnaire
Description: Measure of diabetes self-care. Diabetes Self-Management Questionnaire (DSMQ). 16 items, Scale 0-3. Scoring: Sum and transform to fall between 0-10. Higher score indicates more effective self-care.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
Number analyzed (Participants) | 101 | 99
score on a scale | 8.34 [8.15 to 8.54] | 7.83 [7.63 to 8.03]
Statistical Analysis 1: Comparison: PRACTICE-DM vs Standard VA Home Telehealth; Test type: Equivalence — Difference between groups at 12months; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [0.25 to 0.78]

4. Secondary Outcome: Perceived Competence Scale
Description: Measure of diabetes self-efficacy and capacity. Perceived Competence Scale (PCS). 4 items, Scale 1-7. Scoring: average (1-7) Higher score indicates greater confidence.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
Number analyzed (Participants) | 101 | 99
score on a scale | 6.31 [6.09 to 6.54] | 5.92 [5.69 to 6.16]
Statistical Analysis 1: Comparison: PRACTICE-DM vs Standard VA Home Telehealth; Test type: Equivalence — Difference between groups at 12months; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [0.07 to 0.71]

5. Secondary Outcome: Body Mass Index
Description: Measure of weight at 6months due to low number of 12month in person visits permitting data collection as a result of coronavirus disease 2019 (COVID-19) restrictions
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
Number analyzed (Participants) | 101 | 99
kg/m^2 | 35.05 [34.10 to 36.01] | 34.86 [33.91 to 35.82]
Statistical Analysis 1: Comparison: PRACTICE-DM vs Standard VA Home Telehealth; Test type: Equivalence — Difference between groups at 6months; p = 0.39, Mixed Models Analysis; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.24 to 0.62]

6. Secondary Outcome: Patient Health Questionnaire-8
Description: Measure of depressive symptoms, Patient Health Questionnaire depression scale (PHQ8). 8 items, Scale 0-3, Scoring average of responses 0-24. Higher score indicates greater depressive symptoms.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
Number analyzed (Participants) | 101 | 99
score on a scale | 4.64 [3.62 to 5.66] | 5.80 [4.75 to 6.85]
Statistical Analysis 1: Comparison: PRACTICE-DM vs Standard VA Home Telehealth; Test type: Equivalence — Difference between groups at 12months; p = 0.10, Mixed Models Analysis; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-2.53 to 0.21]

ADVERSE EVENTS:
Time Frame: Adverse events were collected with each patient contact and a systematic review with study outcome visits during the 12month participation.
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Arm/Group | PRACTICE-DM | Standard VA Home Telehealth
All-Cause Mortality (participants affected / at risk) | 0/101 | 1/99
Serious Adverse Events (participants affected / at risk) | 15/101 | 14/99
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRACTICE-DM (N=101) | Standard VA Home Telehealth (N=99)
Hospitalization (Cardiac disorders) | 1 (2) | 1 (1)
Hospitalization (Endocrine disorders) | 2 (3) | 0 (0)
Hospitalization (General disorders) | 0 (0) | 1 (3)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization (Infections and infestations) | 0 (0) | 4 (4)
Hospitalization (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Hospitalization (Immune system disorders) | 1 (1) | 0 (0)
Hospitalization (Nervous system disorders) | 0 (0) | 2 (3)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalization (Psychiatric disorders) | 0 (0) | 2 (2)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Hospitalization (Surgical and medical procedures) | 1 (1) | 2 (2)
Important Medical Event (Cardiac disorders) | 1 (1) | 0 (0)
Important Medical Event (General disorders) | 1 (1) | 0 (0)
Important Medical Event (Infections and infestations) | 1 (1) | 0 (0)
Important Medical Event (Renal and urinary disorders) | 2 (2) | 0 (0)
Important Medical Event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Important Medical Event (Surgical and medical procedures) | 2 (2) | 0 (0)
Persistent or Significant Illness (General disorders) | 1 (1) | 0 (0)
Persistent or Significant Illness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03520413/Prot_SAP_000.pdf